CLINICAL TRIAL: NCT00928876
Title: Effect of Interleukin-1 Receptor Antagonist on Insulin Sensitivity in Obese, Insulin Resistant Individuals
Brief Title: Interleukin-1 Receptor Antagonist and Insulin Sensitivity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Prof. Dr. C.J. Tack, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMCN001
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: anakinra; Diabetes mellitus, type 2; Insulin resistance; Interleukin-1beta
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anakinra group (Experimental): Anakinra 150 mg/day during four weeks
  Interventions: Drug: Anakinra (Kineret)
- Placebo (Placebo Comparator): Placebo during four weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra (Kineret) — anakinra 150 mg s/c. daily for four weeks
  Other Names: kineret
  Arms: Anakinra group
Drug: Placebo — placebo s/c daily for four weeks
  Arms: Placebo

SUMMARY:
Obesity is characterized by continuous low-grade inflammation. This is an important link between obesity and insulin resistance.

Results from the investigators' own group of in vitro and in vivo research on mice show that Interleukin-1 is involved in the process of developing insulin resistance. Earlier it has been shown that interleukin-1 receptor antagonist in human subjects improves glycemic control. The investigators' hypothesis is that this is due to improved insulin sensitivity.

DETAILED DESCRIPTION:
The prevalence of obesity is increasing fast. Obesity is one of the most common acquired risk factors for insulin resistance. As a consequence the prevalence of type 2 diabetes mellitus is rising fast as well.

Interleukin 6 and Tumor Necrosis Factor alfa are well known pro-inflammatory cytokines that have been linked to insulin resistance. Results from our own group show that interleukin-1 is also involved in the process of developing insulin resistance.

Earlier research projects studied the effect of Interleukin-1 receptor antagonist (Anakinra) on glycemic control in subjects with type 2 diabetes mellitus. It was shown that glycemic control was improved. The authors conclude that this is the result of improved function of pancreatic beta cells.

These results are in contrast to our results of in vitro en in vivo research on mice, which show improved insulin sensitivity by Interleukin-1 receptor antagonist.

A possible explanation for not finding an effect on insulin sensitivity by earlier research projects may be that it is difficult to reliable quantify insulin sensitivity in this group of patients with concurrent changes in glycemic control, extensive co-morbidity and medication use, who might be at the rather extreme end of insulin resistance. Furthermore a relatively low dose of Anakinra was used.

Altogether we hypothesize that the effect of Interleukin-1 is not only mediated through better pancreatic beta-cell function, but that Interleukin-1 blocking by recombinant Interleukin-1 receptor antagonist will also diminish insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* adult subjects with a BMI > 30 kg/m2
* 3 or more characteristics of the metabolic syndrome

Exclusion Criteria:

* inability to give informed consent
* age < 18 years
* known diabetes mellitus
* fasting plasma glucose > 7,0 mmol/l or HbA1c > 6,2%
* presence of any medical condition that might interfere with the current study protocol
* immunodeficiency of immunosuppressive treatment
* anti-inflammatory drugs (100 mg of aspirin/day is allowed)
* signs of current infection
* history of recurrent infections
* pregnancy or breast feeding
* liver disease
* renal disease
* neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-03 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
to determine the effect of Interleukin-1 receptor antagonist on insulin sensitivity, as derived from glucose infusion rate measured by euglycemic hyperinsulinemic clamp | after four weeks of treatment

SECONDARY OUTCOMES:
pancreatic beta cell function als tested by oral glucose tolerance test, pro-insulin/insulin ratio | after four weeks of treatment
lipid profile | after four weeks of treatment
systemic inflammation | after four weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: C J Tack, Prof Dr, Study Chair — Radboud University Medical Center
Locations (1):
- Rabdoud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Larsen CM, Faulenbach M, Vaag A, Volund A, Ehses JA, Seifert B, Mandrup-Poulsen T, Donath MY. Interleukin-1-receptor antagonist in type 2 diabetes mellitus. N Engl J Med. 2007 Apr 12;356(15):1517-26. doi: 10.1056/NEJMoa065213. PMID 17429083
- [Derived] van Asseldonk EJ, Stienstra R, Koenen TB, Joosten LA, Netea MG, Tack CJ. Treatment with Anakinra improves disposition index but not insulin sensitivity in nondiabetic subjects with the metabolic syndrome: a randomized, double-blind, placebo-controlled study. J Clin Endocrinol Metab. 2011 Jul;96(7):2119-26. doi: 10.1210/jc.2010-2992. Epub 2011 Apr 20. PMID 21508140